CLINICAL TRIAL: NCT06064669
Title: Effect of Metformin on Healthy Live Birth After In-vitro Fertilization in Women With Prediabetes Mellitus: a Multicenter Double-blind Placebo Controlled Randomized Trial
Brief Title: Effect of Metformin on Healthy Live Birth in Women With Prediabetes
Acronym: MELT-PreDM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University (Other)
Collaborators: Ren Ji Hospital of Shanghai Jiao Tong University (Unknown); Women's Hospital of Zhejiang University (Unknown); Shengjing Hospital (Other); Nanjing Medical University (Other); General Hospital of Ningxia Medical University (Other); West China Second University Hospital (Other); Maternal and Child Health Hospital of Henan Province (Unknown); Qingdao women's and children's Hospital (Unknown)
Responsible Party: Principal Investigator, Chen Zi-Jiang, Academician, Shandong University
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: MELT-PreDM
Record Dates: First submitted 2023-09-19; First posted 2023-10-03 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Metformin; Prediabetes; In-Vitro Fertilization
MeSH Terms: conditions — Prediabetic State

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Metformin-Metformin Group (Experimental): Metformin pretreatment before ovarian stimulation till oocyte retrieval and cryopreservation of all embryos, and followed by metformin pretreatment before endometrial preparation for frozen embryo transfer and till the establishment of clinical pregnancy (7-8 weeks gestation) after the first frozen embryo transfer.
  Interventions: Drug: Metformin pretreatment before ovarian stimulation; Drug: Metformin pretreatment before endometrial preparation for frozen embryo transfer
- Metformin-Placebo Group (Experimental): Metformin pretreatment before ovarian stimulation till oocyte retrieval and cryopreservation of all embryos, and followed by placebo pretreatment before endometrial preparation for frozen embryo transfer and till the establishment of clinical pregnancy (7-8 weeks gestation) after the first frozen embryo transfer.
  Interventions: Drug: Metformin pretreatment before ovarian stimulation; Drug: Placebo pretreatment before endometrial preparation for frozen embryo transfer
- Placebo-Metformin Group (Experimental): Placebo pretreatment before ovarian stimulation till oocyte retrieval and cryopreservation of all embryos, and followed by metformin pretreatment before endometrial preparation for frozen embryo transfer and till the establishment of clinical pregnancy (7-8 weeks gestation) after the first frozen embryo transfer.
  Interventions: Drug: Placebo pretreatment before ovarian stimulation; Drug: Metformin pretreatment before endometrial preparation for frozen embryo transfer
- Placebo-Placebo Group (Experimental): Placebo pretreatment before ovarian stimulation till oocyte retrieval and cryopreservation of all embryos, and followed by placebo pretreatment before endometrial preparation for frozen embryo transfer and till the establishment of clinical pregnancy (7-8 weeks gestation) after the first frozen embryo transfer.
  Interventions: Drug: Placebo pretreatment before ovarian stimulation; Drug: Placebo pretreatment before endometrial preparation for frozen embryo transfer

INTERVENTIONS:
Drug: Metformin pretreatment before ovarian stimulation — The enrolled patients will be prescribed metformin 850mg twice daily for at least 4 weeks prior to ovarian stimulation till oocyte retrieval.
  Other Names: Metformin before ovarian stimulation
  Arms: Metformin-Metformin Group; Metformin-Placebo Group
Drug: Placebo pretreatment before ovarian stimulation — The enrolled patients will be prescribed placebo 850mg twice daily for at least 4 weeks prior to ovarian stimulation till oocyte retrieval.
  Other Names: Placebo before ovarian stimulation
  Arms: Placebo-Metformin Group; Placebo-Placebo Group
Drug: Metformin pretreatment before endometrial preparation for frozen embryo transfer — After oocyte retrieval, the enrolled patients will be prescribed metformin 850mg twice daily for at least 4 weeks before endometrial preparation for frozen embryo transfer and till the establishment of clinical pregnancy (7-8 weeks gestation) after the first frozen embryo transfer.
  Other Names: Metformin before endometrial preparation
  Arms: Metformin-Metformin Group; Placebo-Metformin Group
Drug: Placebo pretreatment before endometrial preparation for frozen embryo transfer — After oocyte retrieval, the enrolled patients will be prescribed placebo 850mg twice daily for at least 4 weeks before endometrial preparation for frozen embryo transfer and till the establishment of clinical pregnancy (7-8 weeks gestation) after the first frozen embryo transfer.
  Other Names: Placebo before endometrial preparation
  Arms: Metformin-Placebo Group; Placebo-Placebo Group

SUMMARY:
To evaluate the efficacy and safety of metformin pretreatment on reproductive outcomes in infertile women with prediabetes.

DETAILED DESCRIPTION:
To evaluate the efficacy and safety of metformin pretreatment on reproductive outcomes in infertile women with prediabetes and to determine whether either starting metformin pretreatment before ovarian stimulation (aiming at improving the quality of oocyte/embryo) or starting before frozen embryo transfer (FET) (aiming at improving the receptivity of endometrium) could increase the chance of a healthy live birth compared with placebo.

ELIGIBILITY:
Inclusion Criteria:

1. Women who are diagnosed with prediabetes by ADA criteria, including either IFG, IGT, or HbA1C 5.7-6.4%.
2. Women aged 20-40 years.
3. Women who plan to undergo a new cycle of IVF, ICSI, or PGT-A.

Exclusion Criteria:

1. Women who are diagnosed with diabetes according to the ADA criteria11,12, which is meeting one of the following criteria: fasting plasma glucose ≥7.0mmol/L, 2-h plasma glucose during 75-g OGTT ≥11.1mmol/L, HbA1c≥6.5%, or a random plasma glucose≥11.1mmol/L.
2. Women who are taking medicine that interfere with glucose metabolism, such as metformin, oral anti-diabetic agents (sulfonylureas, glinides, thiazolidinediones, α-glycosidase inhibitors, GLP-1 receptor agonist, etc.), weight loss drugs (i.e.orlistat, etc.), glucocorticoids, and growth hormones within 2 months before enrollment.
3. Women with un-corrected hyperthyroidism or hypothyroidism.
4. Women with congenital or acquired abnormal uterine cavity including septate uterus, unicornous uterus, uterus duplex, and intrauterine adhesions.
5. Women with a diagnosis of adenomyosis.
6. Women with untreated hydrosalpinx.
7. Women who plan to undergo PGT-SR or PGT-M.
8. Women with major medical comorbidities, such as known liver disease, known renal disease, or known significant anemia.

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 988 (Estimated)
Dates: Start 2024-02-22 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
healthy live birth | From the date of randomization until delivery after the first embryo transfer, up to 16 months
  defined as a singleton live birth at ≥37 weeks, with infant birth weight between 2500 and 4000g and without a major congenital anomaly.

SECONDARY OUTCOMES:
Change in BMI | From the date of randomization until the establishment of clinical pregnancy after the first embryo transfer, up to 26 weeks
  change in body mass index (BMI) from baseline to the establishment of clinical pregnancy.
Change in fasting glucose level | From the date of randomization until the establishment of clinical pregnancy after the first embryo transfer, up to 26 weeks
  change in fasting glucose level from baseline to the establishment of clinical pregnancy.
Change in fasting insulin level | From the date of randomization until the establishment of clinical pregnancy after the first embryo transfer, up to 26 weeks
  change in fasting insulin level from baseline to the establishment of clinical pregnancy.
Change in 2-h levels of glucose after 75-g OGTT | From the date of randomization until the establishment of clinical pregnancy after the first embryo transfer, up to 26 weeks
  change in 2-h levels of glucose after 75-g OGTT from baseline to the establishment of clinical pregnancy.
Change in 2-h levels of insulin after 75-g OGTT | From the date of randomization until the establishment of clinical pregnancy after the first embryo transfer, up to 26 weeks
  change in 2-h levels of insulin after 75-g OGTT from baseline to the establishment of clinical pregnancy.
Days of ovarian stimulation | From the date of randomization until the day of oocyte retrieved, up to 12 weeks
  the duration of ovarian stimulation by exogenous gonadotropin
Total dose of gonadotropins | From the date of randomization until the day of oocyte retrieved, up to 12 weeks
  the total dose of exogenous gonadotropin used during ovarian stimulation
Peak estradiol level | From the date of randomization until the day of oocyte retrieved, up to 12 weeks
  the estradiol level on the day of hCG trigger
Number of oocyte retrieved | From the date of randomization until the day of oocyte retrieved, up to 12 weeks
  the number of oocyte retrieved
Number of good-score embryos | From the date of randomization until the third day after oocyte retrieval, up to 12 weeks
  the number of good-score embryos
Number of euploid embryos | From the date of randomization until the initiation of endometrial preparation for frozen embryo transfer, up to 20 weeks
  the number of euploid embryos
OHSS | From the day of oocyte retrieved until the initiation of endometrial preparation for the first frozen embryo transfer, up to 8 weeks
  ovarian hyperstimulation syndrome was defined according to the Golan criteria
Clinical pregnancy | 30-35 days after the first frozen embryo transfer
  defined as the ultrasound confirmation of at least one intrauterine gestational sac
Singleton or twin pregnancy | 30-35 days after the first frozen embryo transfer
  the number of intrauterine gestational sacs
Pregnancy loss | From the date of confirmation of pregnancy until the date of pregnancy loss, up to 9 months
  defined as pregnancies that eventuate in a spontaneous abortion or therapeutic abortion that occurred throughout pregnancy.
Live birth | From the date of randomization until delivery after the first embryo transfer, up to 16 months
  defined as the delivery of any neonate with signs of life at ≥ 28 weeks of gestation
Incidences of obstetric and neonatal complications | From the establishment of clinically recognized pregnancy until six weeks after delivery after the first embryo transfer, up to 11 months
  including gestational diabetes mellitus, pre-eclampsia, premature rupture of membrane, placenta previa, placental abruption, congenital anomalies, postpartum hemorrhage, stillbirth, neonatal respiratory distress syndrome, neonatal jaundice, neonatal infection, neonatal death.
Gestational weight gain | at delivery
  maternal weight gain during pregnancy
Birth weight | at delivery
  birth weight of the newborn at delivery
LGA | at delivery
  defined as the birthweight above the 90th percentile for gestational age based on a sex-specific reference
SGA | at delivery
  defined as the birthweight below the 10th percentile for gestational age based on a sex-specific reference
LBW | at delivery
  the infant born weighing less than 2500g
Macrosomia | at delivery
  the infant born weighing larger than 4000g
Adverse events | From the date of randomization until six weeks after delivery after the first embryo transfer, up to 18 months
  adverse event (AE) and serious adverse event (SAE)
Cumulative live birth | From the date of randomization until delivery, up to 28 months
  define as women achieving live birth after all the cycles of embryo transfer per oocyte retrieval that performed within one year after randomization.

CONTACTS AND LOCATIONS:
Overall Officials: Zi-Jiang Chen, Professor, Principal Investigator — Shandong University
Locations (1):
- Shandong University, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Yes
Deidentified participant data
Supporting Information: Study Protocol, SAP
Time Frame: 6 months after publication
Access Criteria: The data of this study are available on request from the corresponding author

REFERENCES:
- [Background] Wei Y, Xu Q, Yang H, Yang Y, Wang L, Chen H, Anderson C, Liu X, Song G, Li Q, Wang Q, Shen H, Zhang Y, Yan D, Peng Z, He Y, Wang Y, Zhang Y, Zhang H, Ma X. Preconception diabetes mellitus and adverse pregnancy outcomes in over 6.4 million women: A population-based cohort study in China. PLoS Med. 2019 Oct 1;16(10):e1002926. doi: 10.1371/journal.pmed.1002926. eCollection 2019 Oct. PMID 31574092
- [Background] Macintosh MC, Fleming KM, Bailey JA, Doyle P, Modder J, Acolet D, Golightly S, Miller A. Perinatal mortality and congenital anomalies in babies of women with type 1 or type 2 diabetes in England, Wales, and Northern Ireland: population based study. BMJ. 2006 Jul 22;333(7560):177. doi: 10.1136/bmj.38856.692986.AE. Epub 2006 Jun 16. PMID 16782722
- [Background] Egan AM, Dow ML, Vella A. A Review of the Pathophysiology and Management of Diabetes in Pregnancy. Mayo Clin Proc. 2020 Dec;95(12):2734-2746. doi: 10.1016/j.mayocp.2020.02.019. Epub 2020 Jul 28. PMID 32736942
- [Background] Bianco ME, Josefson JL. Hyperglycemia During Pregnancy and Long-Term Offspring Outcomes. Curr Diab Rep. 2019 Nov 21;19(12):143. doi: 10.1007/s11892-019-1267-6. PMID 31754898
- [Background] Farrar D, Simmonds M, Bryant M, Sheldon TA, Tuffnell D, Golder S, Dunne F, Lawlor DA. Hyperglycaemia and risk of adverse perinatal outcomes: systematic review and meta-analysis. BMJ. 2016 Sep 13;354:i4694. doi: 10.1136/bmj.i4694. PMID 27624087
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Armengaud JB, Ma RCW, Siddeek B, Visser GHA, Simeoni U. Offspring of mothers with hyperglycaemia in pregnancy: The short term and long-term impact. What is new? Diabetes Res Clin Pract. 2018 Nov;145:155-166. doi: 10.1016/j.diabres.2018.07.039. Epub 2018 Aug 6. PMID 30092235
- [Background] Kitzmiller JL, Buchanan TA, Kjos S, Combs CA, Ratner RE. Pre-conception care of diabetes, congenital malformations, and spontaneous abortions. Diabetes Care. 1996 May;19(5):514-41. doi: 10.2337/diacare.19.5.514. No abstract available. PMID 8732721
- [Background] Correa A, Gilboa SM, Besser LM, Botto LD, Moore CA, Hobbs CA, Cleves MA, Riehle-Colarusso TJ, Waller DK, Reece EA. Diabetes mellitus and birth defects. Am J Obstet Gynecol. 2008 Sep;199(3):237.e1-9. doi: 10.1016/j.ajog.2008.06.028. Epub 2008 Jul 31. PMID 18674752
- [Background] Faerch K, Vaag A, Holst JJ, Hansen T, Jorgensen T, Borch-Johnsen K. Natural history of insulin sensitivity and insulin secretion in the progression from normal glucose tolerance to impaired fasting glycemia and impaired glucose tolerance: the Inter99 study. Diabetes Care. 2009 Mar;32(3):439-44. doi: 10.2337/dc08-1195. Epub 2008 Dec 3. PMID 19056613
- [Background] Li R, Wu J, He J, Wang Y, Liu X, Chen X, Tong C, Ding Y, Su Y, Chen W, Zhang C, Gao R. Mice endometrium receptivity in early pregnancy is impaired by maternal hyperinsulinemia. Mol Med Rep. 2017 May;15(5):2503-2510. doi: 10.3892/mmr.2017.6322. Epub 2017 Mar 14. PMID 28447735
- [Background] Chang EM, Han JE, Seok HH, Lee DR, Yoon TK, Lee WS. Insulin resistance does not affect early embryo development but lowers implantation rate in in vitro maturation-in vitro fertilization-embryo transfer cycle. Clin Endocrinol (Oxf). 2013 Jul;79(1):93-9. doi: 10.1111/cen.12099. Epub 2013 Apr 19. PMID 23176069
- [Background] Via Y Rada R, Daniel N, Archilla C, Frambourg A, Jouneau L, Jaszczyszyn Y, Charpigny G, Duranthon V, Calderari S. Identification of the Inner Cell Mass and the Trophectoderm Responses after an In Vitro Exposure to Glucose and Insulin during the Preimplantation Period in the Rabbit Embryo. Cells. 2022 Nov 25;11(23):3766. doi: 10.3390/cells11233766. PMID 36497026
- [Background] Jungheim ES, Moley KH. The impact of type 1 and type 2 diabetes mellitus on the oocyte and the preimplantation embryo. Semin Reprod Med. 2008 Mar;26(2):186-95. doi: 10.1055/s-2008-1042957. PMID 18302110
- [Background] Catalano PM, Shankar K. Obesity and pregnancy: mechanisms of short term and long term adverse consequences for mother and child. BMJ. 2017 Feb 8;356:j1. doi: 10.1136/bmj.j1. PMID 28179267
- [Background] Coussa A, Hasan HA, Barber TM. Effects of in vitro fertilization (IVF) therapies on metabolic, endocrine and inflammatory status in IVF-conceived pregnancy. Clin Endocrinol (Oxf). 2020 Dec;93(6):705-712. doi: 10.1111/cen.14270. Epub 2020 Jul 9. PMID 32578220
- [Background] Coussa A, Hasan HA, Barber TM. Impact of contraception and IVF hormones on metabolic, endocrine, and inflammatory status. J Assist Reprod Genet. 2020 Jun;37(6):1267-1272. doi: 10.1007/s10815-020-01756-z. Epub 2020 Mar 25. PMID 32215823
- [Background] Wei D, Zhang B, Shi Y, Zhang L, Zhao S, Du Y, Xu L, Legro RS, Zhang H, Chen ZJ. Effect of Preconception Impaired Glucose Tolerance on Pregnancy Outcomes in Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2017 Oct 1;102(10):3822-3829. doi: 10.1210/jc.2017-01294. PMID 28938429
- [Background] Wang W, Tang X, Jiang Q, Niu Y, Wang Z, Wei D. Risk factors for clinical pregnancy loss after IVF in women with PCOS. Reprod Biomed Online. 2023 Jan;46(1):107-114. doi: 10.1016/j.rbmo.2022.10.002. Epub 2022 Oct 12. PMID 36396532
- [Background] Christ JP, Gunning MN, Meun C, Eijkemans MJC, van Rijn BB, Bonsel GJ, Laven JSE, Fauser BCJM. Pre-Conception Characteristics Predict Obstetrical and Neonatal Outcomes in Women With Polycystic Ovary Syndrome. J Clin Endocrinol Metab. 2019 Mar 1;104(3):809-818. doi: 10.1210/jc.2018-01787. PMID 30590587
- [Background] Wei HJ, Young R, Kuo IL, Liaw CM, Chiang HS, Yeh CY. Abnormal preconception oral glucose tolerance test predicts an unfavorable pregnancy outcome after an in vitro fertilization cycle. Fertil Steril. 2008 Sep;90(3):613-8. doi: 10.1016/j.fertnstert.2007.07.1289. Epub 2007 Nov 5. PMID 17980878
- [Background] Lao TT, Ho LF. Impaired glucose tolerance and pregnancy outcome in Chinese women with high body mass index. Hum Reprod. 2000 Aug;15(8):1826-9. doi: 10.1093/humrep/15.8.1826. PMID 10920111
- [Background] Zolghadri J, Tavana Z, Kazerooni T, Soveid M, Taghieh M. Relationship between abnormal glucose tolerance test and history of previous recurrent miscarriages, and beneficial effect of metformin in these patients: a prospective clinical study. Fertil Steril. 2008 Sep;90(3):727-30. doi: 10.1016/j.fertnstert.2007.06.079. Epub 2007 Nov 14. PMID 18001723
- [Background] Cho NH, Shaw JE, Karuranga S, Huang Y, da Rocha Fernandes JD, Ohlrogge AW, Malanda B. IDF Diabetes Atlas: Global estimates of diabetes prevalence for 2017 and projections for 2045. Diabetes Res Clin Pract. 2018 Apr;138:271-281. doi: 10.1016/j.diabres.2018.02.023. Epub 2018 Feb 26. PMID 29496507
- [Background] Nanditha A, Ma RC, Ramachandran A, Snehalatha C, Chan JC, Chia KS, Shaw JE, Zimmet PZ. Diabetes in Asia and the Pacific: Implications for the Global Epidemic. Diabetes Care. 2016 Mar;39(3):472-85. doi: 10.2337/dc15-1536. PMID 26908931
- [Background] Legro RS, Gnatuk CL, Kunselman AR, Dunaif A. Changes in glucose tolerance over time in women with polycystic ovary syndrome: a controlled study. J Clin Endocrinol Metab. 2005 Jun;90(6):3236-42. doi: 10.1210/jc.2004-1843. Epub 2005 Mar 29. PMID 15797965
- [Background] Legro RS, Arslanian SA, Ehrmann DA, Hoeger KM, Murad MH, Pasquali R, Welt CK; Endocrine Society. Diagnosis and treatment of polycystic ovary syndrome: an Endocrine Society clinical practice guideline. J Clin Endocrinol Metab. 2013 Dec;98(12):4565-92. doi: 10.1210/jc.2013-2350. Epub 2013 Oct 22. PMID 24151290
- [Background] Wahabi HA, Fayed A, Esmaeil S, Elmorshedy H, Titi MA, Amer YS, Alzeidan RA, Alodhayani AA, Saeed E, Bahkali KH, Kahili-Heede MK, Jamal A, Sabr Y. Systematic review and meta-analysis of the effectiveness of pre-pregnancy care for women with diabetes for improving maternal and perinatal outcomes. PLoS One. 2020 Aug 18;15(8):e0237571. doi: 10.1371/journal.pone.0237571. eCollection 2020. PMID 32810195
- [Background] Glinianaia SV, Tennant PW, Crowder D, Nayar R, Bell R. Fifteen-year trends and predictors of preparation for pregnancy in women with pre-conception Type 1 and Type 2 diabetes: a population-based cohort study. Diabet Med. 2014 Sep;31(9):1104-13. doi: 10.1111/dme.12460. Epub 2014 Apr 21. PMID 24702102
- [Background] American College of Obstetricians and Gynecologists' Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 201: Pregestational Diabetes Mellitus. Obstet Gynecol. 2018 Dec;132(6):e228-e248. doi: 10.1097/AOG.0000000000002960. PMID 30461693
- [Background] Pan XR, Li GW, Hu YH, Wang JX, Yang WY, An ZX, Hu ZX, Lin J, Xiao JZ, Cao HB, Liu PA, Jiang XG, Jiang YY, Wang JP, Zheng H, Zhang H, Bennett PH, Howard BV. Effects of diet and exercise in preventing NIDDM in people with impaired glucose tolerance. The Da Qing IGT and Diabetes Study. Diabetes Care. 1997 Apr;20(4):537-44. doi: 10.2337/diacare.20.4.537. PMID 9096977
- [Background] Tuomilehto J, Lindstrom J, Eriksson JG, Valle TT, Hamalainen H, Ilanne-Parikka P, Keinanen-Kiukaanniemi S, Laakso M, Louheranta A, Rastas M, Salminen V, Uusitupa M; Finnish Diabetes Prevention Study Group. Prevention of type 2 diabetes mellitus by changes in lifestyle among subjects with impaired glucose tolerance. N Engl J Med. 2001 May 3;344(18):1343-50. doi: 10.1056/NEJM200105033441801. PMID 11333990
- [Background] Knowler WC, Barrett-Connor E, Fowler SE, Hamman RF, Lachin JM, Walker EA, Nathan DM; Diabetes Prevention Program Research Group. Reduction in the incidence of type 2 diabetes with lifestyle intervention or metformin. N Engl J Med. 2002 Feb 7;346(6):393-403. doi: 10.1056/NEJMoa012512. PMID 11832527
- [Background] Galaviz KI, Weber MB, Suvada K BS, Gujral UP, Wei J, Merchant R, Dharanendra S, Haw JS, Narayan KMV, Ali MK. Interventions for Reversing Prediabetes: A Systematic Review and Meta-Analysis. Am J Prev Med. 2022 Apr;62(4):614-625. doi: 10.1016/j.amepre.2021.10.020. Epub 2022 Feb 10. PMID 35151523
- [Background] Hostalek U, Campbell I. Metformin for diabetes prevention: update of the evidence base. Curr Med Res Opin. 2021 Oct;37(10):1705-1717. doi: 10.1080/03007995.2021.1955667. Epub 2021 Jul 28. PMID 34281467
- [Background] Ratner RE, Christophi CA, Metzger BE, Dabelea D, Bennett PH, Pi-Sunyer X, Fowler S, Kahn SE; Diabetes Prevention Program Research Group. Prevention of diabetes in women with a history of gestational diabetes: effects of metformin and lifestyle interventions. J Clin Endocrinol Metab. 2008 Dec;93(12):4774-9. doi: 10.1210/jc.2008-0772. Epub 2008 Sep 30. PMID 18826999
- [Background] Rowan JA, Hague WM, Gao W, Battin MR, Moore MP; MiG Trial Investigators. Metformin versus insulin for the treatment of gestational diabetes. N Engl J Med. 2008 May 8;358(19):2003-15. doi: 10.1056/NEJMoa0707193. PMID 18463376
- [Background] Lovvik TS, Carlsen SM, Salvesen O, Steffensen B, Bixo M, Gomez-Real F, Lonnebotn M, Hestvold KV, Zabielska R, Hirschberg AL, Trouva A, Thorarinsdottir S, Hjelle S, Berg AH, Andrae F, Poromaa IS, Mohlin J, Underdal M, Vanky E. Use of metformin to treat pregnant women with polycystic ovary syndrome (PregMet2): a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2019 Apr;7(4):256-266. doi: 10.1016/S2213-8587(19)30002-6. Epub 2019 Feb 18. PMID 30792154
- [Background] Chiswick C, Reynolds RM, Denison F, Drake AJ, Forbes S, Newby DE, Walker BR, Quenby S, Wray S, Weeks A, Lashen H, Rodriguez A, Murray G, Whyte S, Norman JE. Effect of metformin on maternal and fetal outcomes in obese pregnant women (EMPOWaR): a randomised, double-blind, placebo-controlled trial. Lancet Diabetes Endocrinol. 2015 Oct;3(10):778-86. doi: 10.1016/S2213-8587(15)00219-3. Epub 2015 Jul 9. PMID 26165398
- [Background] Tieu J, Coat S, Hague W, Middleton P, Shepherd E. Oral anti-diabetic agents for women with established diabetes/impaired glucose tolerance or previous gestational diabetes planning pregnancy, or pregnant women with pre-existing diabetes. Cochrane Database Syst Rev. 2017 Oct 18;10(10):CD007724. doi: 10.1002/14651858.CD007724.pub3. PMID 29045765
- [Background] Kovo M, Haroutiunian S, Feldman N, Hoffman A, Glezerman M. Determination of metformin transfer across the human placenta using a dually perfused ex vivo placental cotyledon model. Eur J Obstet Gynecol Reprod Biol. 2008 Jan;136(1):29-33. doi: 10.1016/j.ejogrb.2007.01.013. Epub 2007 Mar 12. PMID 17350747
- [Background] Sharpe A, Morley LC, Tang T, Norman RJ, Balen AH. Metformin for ovulation induction (excluding gonadotrophins) in women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2019 Dec 17;12(12):CD013505. doi: 10.1002/14651858.CD013505. PMID 31845767
- [Background] Tso LO, Costello MF, Albuquerque LET, Andriolo RB, Macedo CR. Metformin treatment before and during IVF or ICSI in women with polycystic ovary syndrome. Cochrane Database Syst Rev. 2020 Dec 21;12(12):CD006105. doi: 10.1002/14651858.CD006105.pub4. PMID 33347618
- [Background] Wu Y, Tu M, Huang Y, Liu Y, Zhang D. Association of Metformin With Pregnancy Outcomes in Women With Polycystic Ovarian Syndrome Undergoing In Vitro Fertilization: A Systematic Review and Meta-analysis. JAMA Netw Open. 2020 Aug 3;3(8):e2011995. doi: 10.1001/jamanetworkopen.2020.11995. PMID 32744629
- [Background] Picon-Cesar MJ, Molina-Vega M, Suarez-Arana M, Gonzalez-Mesa E, Sola-Moyano AP, Roldan-Lopez R, Romero-Narbona F, Olveira G, Tinahones FJ, Gonzalez-Romero S. Metformin for gestational diabetes study: metformin vs insulin in gestational diabetes: glycemic control and obstetrical and perinatal outcomes: randomized prospective trial. Am J Obstet Gynecol. 2021 Nov;225(5):517.e1-517.e17. doi: 10.1016/j.ajog.2021.04.229. Epub 2021 Apr 19. PMID 33887240
- [Background] Balsells M, Garcia-Patterson A, Sola I, Roque M, Gich I, Corcoy R. Glibenclamide, metformin, and insulin for the treatment of gestational diabetes: a systematic review and meta-analysis. BMJ. 2015 Jan 21;350:h102. doi: 10.1136/bmj.h102. PMID 25609400
- [Background] Abolhassani N, Winterfeld U, Kaplan YC, Jaques C, Minder Wyssmann B, Del Giovane C, Panchaud A. Major malformations risk following early pregnancy exposure to metformin: a systematic review and meta-analysis. BMJ Open Diabetes Res Care. 2023 Jan;11(1):e002919. doi: 10.1136/bmjdrc-2022-002919. PMID 36720508
- [Background] Glueck CJ, Goldenberg N, Pranikoff J, Loftspring M, Sieve L, Wang P. Height, weight, and motor-social development during the first 18 months of life in 126 infants born to 109 mothers with polycystic ovary syndrome who conceived on and continued metformin through pregnancy. Hum Reprod. 2004 Jun;19(6):1323-30. doi: 10.1093/humrep/deh263. Epub 2004 Apr 29. PMID 15117896
- [Background] Bordewijk EM, Nahuis M, Costello MF, Van der Veen F, Tso LO, Mol BW, van Wely M. Metformin during ovulation induction with gonadotrophins followed by timed intercourse or intrauterine insemination for subfertility associated with polycystic ovary syndrome. Cochrane Database Syst Rev. 2017 Jan 24;1(1):CD009090. doi: 10.1002/14651858.CD009090.pub2. PMID 28118681
- [Background] Unanyan A, Pivazyan L, Krylova E, Eskin A, Zakaryan A, Sarkisova A, Ishchenko A. Effectiveness of inositol, metformin and their combination in women with PCOS undergoing assisted reproduction: systematic review and meta-analysis. Gynecol Endocrinol. 2022 Dec;38(12):1035-1046. doi: 10.1080/09513590.2022.2136160. Epub 2022 Oct 26. PMID 36285403
- [Background] Ryssdal M, Vanky E, Stokkeland LMT, Jarmund AH, Steinkjer B, Lovvik TS, Madssen TS, Iversen AC, Giskeodegard GF. Immunomodulatory Effects of Metformin Treatment in Pregnant Women With PCOS. J Clin Endocrinol Metab. 2023 Aug 18;108(9):e743-e753. doi: 10.1210/clinem/dgad145. PMID 36916886
- [Background] Beyuo T, Obed SA, Adjepong-Yamoah KK, Bugyei KA, Oppong SA, Marfoh K. Metformin versus Insulin in the Management of Pre-Gestational Diabetes Mellitus in Pregnancy and Gestational Diabetes Mellitus at the Korle Bu Teaching Hospital: A Randomized Clinical Trial. PLoS One. 2015 May 6;10(5):e0125712. doi: 10.1371/journal.pone.0125712. eCollection 2015. PMID 25945500
- [Background] Legro RS. Metformin as adjuvant therapy to IVF in women with PCOS: when is intention-to-treat unintentional? Hum Reprod. 2011 Aug;26(8):2043-4. doi: 10.1093/humrep/der155. Epub 2011 May 23. No abstract available. PMID 21606132
- [Background] American Diabetes Association. Diagnosis and classification of diabetes mellitus. Diabetes Care. 2014 Jan;37 Suppl 1:S81-90. doi: 10.2337/dc14-S081. No abstract available. PMID 24357215
- [Background] ElSayed NA, Aleppo G, Aroda VR, Bannuru RR, Brown FM, Bruemmer D, Collins BS, Hilliard ME, Isaacs D, Johnson EL, Kahan S, Khunti K, Leon J, Lyons SK, Perry ML, Prahalad P, Pratley RE, Seley JJ, Stanton RC, Gabbay RA, on behalf of the American Diabetes Association. 2. Classification and Diagnosis of Diabetes: Standards of Care in Diabetes-2023. Diabetes Care. 2023 Jan 1;46(Suppl 1):S19-S40. doi: 10.2337/dc23-S002. PMID 36507649
- [Background] Wei D, Liu JY, Sun Y, Shi Y, Zhang B, Liu JQ, Tan J, Liang X, Cao Y, Wang Z, Qin Y, Zhao H, Zhou Y, Ren H, Hao G, Ling X, Zhao J, Zhang Y, Qi X, Zhang L, Deng X, Chen X, Zhu Y, Wang X, Tian LF, Lv Q, Ma X, Zhang H, Legro RS, Chen ZJ. Frozen versus fresh single blastocyst transfer in ovulatory women: a multicentre, randomised controlled trial. Lancet. 2019 Mar 30;393(10178):1310-1318. doi: 10.1016/S0140-6736(18)32843-5. Epub 2019 Feb 28. PMID 30827784
- [Background] Zuo N, Gao Y, Zhang N, Li D, Wang X. Effects of immediate versus delayed frozen embryo transfer in high responder patients undergoing freeze-all cycles. BMC Pregnancy Childbirth. 2021 Jun 28;21(1):455. doi: 10.1186/s12884-021-03919-x. PMID 34182954
- [Background] Huang J, Lin J, Lu X, Cai R, Song N, Kuang Y. Delayed versus immediate frozen embryo transfer after oocyte retrieval: a systematic review and meta-analysis. J Assist Reprod Genet. 2020 Aug;37(8):1949-1957. doi: 10.1007/s10815-020-01857-9. Epub 2020 Jun 19. PMID 32556707
- [Background] Yildiz S, Turkgeldi E, Kalafat E, Keles I, Gokyer D, Ata B. Do live birth rate and obstetric outcomes vary between immediate and delayed embryo transfers following freeze-all cycles? J Gynecol Obstet Hum Reprod. 2021 Dec;50(10):102224. doi: 10.1016/j.jogoh.2021.102224. Epub 2021 Sep 8. PMID 34506996
- [Background] Lattes K, Checa MA, Vassena R, Brassesco M, Vernaeve V. There is no evidence that the time from egg retrieval to embryo transfer affects live birth rates in a freeze-all strategy. Hum Reprod. 2017 Feb;32(2):368-374. doi: 10.1093/humrep/dew306. Epub 2016 Dec 16. PMID 27986819
- [Background] Santos-Ribeiro S, Siffain J, Polyzos NP, van de Vijver A, van Landuyt L, Stoop D, Tournaye H, Blockeel C. To delay or not to delay a frozen embryo transfer after a failed fresh embryo transfer attempt? Fertil Steril. 2016 May;105(5):1202-1207.e1. doi: 10.1016/j.fertnstert.2015.12.140. Epub 2016 Jan 21. PMID 26806686
- [Background] Santos-Ribeiro S, Polyzos NP, Lan VT, Siffain J, Mackens S, Van Landuyt L, Tournaye H, Blockeel C. The effect of an immediate frozen embryo transfer following a freeze-all protocol: a retrospective analysis from two centres. Hum Reprod. 2016 Nov;31(11):2541-2548. doi: 10.1093/humrep/dew194. Epub 2016 Sep 8. PMID 27609984
- [Background] Song JY, Dong FY, Li L, Zhang XX, Wang AJ, Zhang Y, Gao DD, Xiao JM, Sun ZG. Immediate versus delayed frozen embryo transfer in women following a failed IVF-ET attempt: a multicenter randomized controlled trial. Reprod Biol Endocrinol. 2021 Aug 30;19(1):131. doi: 10.1186/s12958-021-00819-9. PMID 34461950
- [Background] Li H, Sun X, Yang J, Li L, Zhang W, Lu X, Chen J, Chen H, Yu M, Fu W, Peng X, Chen J, Ng EHY. Immediate versus delayed frozen embryo transfer in patients following a stimulated IVF cycle: a randomised controlled trial. Hum Reprod. 2021 Jun 18;36(7):1832-1840. doi: 10.1093/humrep/deab071. PMID 33885131
- [Background] Practice Committee of the American Society for Reproductive Medicine and the Practice Committee for the Society for Assisted Reproductive Technologies. Electronic address: ASRM@asrm.org. Guidance on the limits to the number of embryos to transfer: a committee opinion. Fertil Steril. 2021 Sep;116(3):651-654. doi: 10.1016/j.fertnstert.2021.06.050. Epub 2021 Jul 28. PMID 34330423
- [Background] Wei D, Sun Y, Liu J, Liang X, Zhu Y, Shi Y, Chen ZJ. Live birth after fresh versus frozen single blastocyst transfer (Frefro-blastocyst): study protocol for a randomized controlled trial. Trials. 2017 Jun 5;18(1):253. doi: 10.1186/s13063-017-1993-5. PMID 28583140